CLINICAL TRIAL: NCT01825889
Title: Pharmacokinetics of Evacetrapib (LY2484595) Following Administration to Subjects With Impaired Renal Function
Brief Title: A Study of Evacetrapib (LY2484595) in Participants With Severe Renal Impairment and in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14620; I1V-MC-EIAR (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-02

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — evacetrapib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evacetrapib (Participants With Renal Impairment) (Experimental): Single oral dose of 130 milligrams (mg) evacetrapib on Day 1 to participants with severe renal impairment.
  Interventions: Drug: Evacetrapib
- Evacetrapib (Healthy Participants) (Experimental): Single oral dose of 130 mg evacetrapib on Day 1 to participants with normal renal function.
  Interventions: Drug: Evacetrapib

INTERVENTIONS:
Drug: Evacetrapib
  Other Names: LY2484595

SUMMARY:
The purpose of this study is to measure how much of the study drug, evacetrapib, enters the blood stream and how long it takes the body to dispose of the study drug when given to participants with severe renal (kidney) impairment compared to participants with normal renal (kidney) function. This study will last approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female participants are not of child-bearing potential
* Have a body mass index of 18 to 40 kilograms per square meter (kg/m^2)
* Participants with normal renal function - healthy as determined by medical history, physical examination, and other screening procedures, with normal renal function (assessed by estimated creatinine clearance [CLcr] greater than or equal to 90 milliliters per minute [mL/min] at screening)
* Participants with severe renal impairment - estimated CLcr less than 30 mL/min at screening and are not undergoing hemodialysis

Exclusion Criteria:

* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Participants who are unwilling to comply with the dietary requirements/restrictions during the study
* Hemoglobin less than 9 grams/deciliter (g/dL) or significant active hematological disease from causes other than underlying renal disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Paul, Minnesota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Evacetrapib (Participants With Renal Impairment) | Evacetrapib (Healthy Participants)
Started | 10 | 10
Received One Dose of Study Drug | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Evacetrapib (Participants With Renal Impairment): Single oral dose of 130 mg evacetrapib on Day 1 to participants with severe renal impairment.
- Total: Total of all reporting groups
Arm/Group | Evacetrapib (Participants With Renal Impairment) | Evacetrapib (Healthy Participants) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (9.6) | 61.5 (8.0) | 63.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 6 | 9 | 15
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under The Concentration Versus Time Curve From Time Zero To Time Tlast, Where Tlast is the Last Time Point With a Measurable Concentration (AUC[0-Tlast]) of Evacetrapib
Time Frame: Predose and 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, 264, 312, and 336 hours postdose
Population: All participants who received evacetrapib and had evaluable AUC(0-Tlast) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*h/mL)
Arm/Group | Evacetrapib (Participants With Renal Impairment) | Evacetrapib (Healthy Participants)
Number analyzed (Participants) | 10 | 10
nanograms*hours/milliliter (ng*h/mL) | 15200 (49) | 16000 (37)

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve From Time Zero to Infinity (AUC[0-∞]) of Evacetrapib
Time Frame: Predose and 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, 264, 312, and 336 hours postdose
Population: All participants who received evacetrapib and had evaluable AUC(0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Evacetrapib (Participants With Renal Impairment) | Evacetrapib (Healthy Participants)
Number analyzed (Participants) | 10 | 10
ng*h/mL | 15500 (50) | 16300 (39)

3. Secondary Outcome: Pharmacokinetics (PK): Observed Maximum Concentration (Cmax) of Evacetrapib
Time Frame: Predose and 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, 264, 312, and 336 hours postdose
Population: All participants who received evacetrapib and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Evacetrapib (Participants With Renal Impairment) | Evacetrapib (Healthy Participants)
Number analyzed (Participants) | 10 | 10
nanograms/milliliter (ng/mL) | 969 (43) | 1140 (44)

ADVERSE EVENTS:
Arm/Group | Evacetrapib (Participants With Renal Impairment) | Evacetrapib (Healthy Participants)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evacetrapib (Participants With Renal Impairment) (N=10) | Evacetrapib (Healthy Participants) (N=10)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1)
Vessel puncture site swelling (General disorders) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days